CLINICAL TRIAL: NCT01480778
Title: Pharmacodynamic Assessment to Drug Ciclo 21 (Levonorgestrel + Ethinyl Estradiol) Market by União Química Farmacêutica Nacional S/A Compared to Drug Nordette of Wieth Indústria Farmacêutica Ltda.
Brief Title: Evaluation of Ciclo 21® Effect (Levonorgestrel + Ethinyl Estradiol) Compared to Nordette®.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azidus Brasil (Industry)
Collaborators: União Química Farmacêutica Nacional S/A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LEEUNI0811
Record Dates: First submitted 2011-11-25; First posted 2011-11-29 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Irregular Periods
Keywords: hormonal response, levonorgestrel, ethinyl estradiol
MeSH Terms: conditions — Menstruation Disturbances | interventions — Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LNG+EE2 (Experimental): pill test contained levonorgestrel 0,15 mg and ethynil estradiol 0,03 mg per day over 21 days
  Interventions: Drug: LNG+EE2
- Nordette (Active Comparator): pill comparator contained levonorgestrel 0,15 mg and ethynil estradiol 0,03 mg per day over 21 days
  Interventions: Drug: Nordette

INTERVENTIONS:
Drug: LNG+EE2 — Administration of one pill contained 0.15 mg of levonosgestrel and 0.03 mg of ethynil estradiol per day over 21 days.
  Other Names: Ciclo 21
  Arms: LNG+EE2
Drug: Nordette — Administration of one pill contained 0.15 mg of levonosgestrel and 0.03 mg of ethynil estradiol per day over 21 days.
  Other Names: LNG+EE2
  Arms: Nordette

SUMMARY:
Assessment of the pharmacodynamic profile of the drug Ciclo 21 ®, marketed by União Química Farmacêutica Nacional S / A, compared to the drug Nordette ® Laboratory Wyeth Pharmaceutical Ltda. Through the modulation of hormonal response (inhibition of the pituitary) evidenced by measurement serum LH and FSH for 28 days, as well as by the absence of follicle formation demonstrated by transvaginal ultrasound examinations

DETAILED DESCRIPTION:
secondary objective

* Evaluation of the safety aspects of medicines such as type, frequency and intensity of adverse events between groups during the 28 day trial.

exploratory objective

* Evaluation of the pharmacokinetics of the drug administered through the dosage of serum hormone levonorgestrel and ethinyl estradiol for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Comply with all study procedures, sign, initial and date back, of their own free will, the IC;
2. Women aged between 18 and 35 years, regardless of race and class;
3. Make use of safe non-hormonal method of contraception such as tubal ligation, non-hormonal IUDs or condoms, or be hysterectomised or be vasectomized sexual partner;
4. Examination of Beta-HCG negative;
5. with regular menstrual cycles every 24 to 32 days, at least the last three months;
6. present normal Pap test (current or during the past 02 years);
7. Present or vaginal examination found that the changes do not interfere in the study;
8. present levels of FSH, LH, estradiol and TT for the normal menstrual cycle, as well as normal transvaginal sonographic reports.

Exclusion Criteria:

1. Provide a contraindication to the use of steroids;
2. Use regular or prediction of drugs that interfere with the metabolism of the investigational products, such as antibiotics, anticonvulsants, anticoagulants and hypoglycemic drugs;
3. smokers or have stopped smoking less than 12 months;
4. Diabetic;
5. Toxic-dependent;
6. BMI <18 and> 25;
7. have made use of topical or systemic sex hormone for at least two months before the start of the study;
8. Background and personal or family history of thrombosis or bleeding disorders or vascular disorders or cardiovascular disease;
9. Laboratory tests, gynecological ultrasound or changed, the medical criteria;
10. Individuals with allergies or rheumatic diseases for which is indicated the use of cortico-steroid medication;
11. carry any endocrine changes, especially pituitary and gonadal and / or who are advised to use hormones;
12. with lesions or abnormalities suspected or confirmed in the gonads.
13. personal or family history of breast cancer or other hormone-dependent breast pathology;
14. with hypertension or diabetes mellitus (for drug interactions between the COC and hypoglycemic agents and antihypertensives);

a) History of nausea with oral use of COCs; p) Any condition that may interfere with the discretion of the investigator in the study data as well as being the measurement of the study be deleterious to the patient.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the changes in FSH and LH secretion induced by daily administration of the drug for 21 consecutive days during the 28 days of participation in the trial. | 1, 2, 4, 7, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 24 and 28 days

SECONDARY OUTCOMES:
Safety of drugs: type, frequency and intensity of adverse events between groups during the 28 day trial. Exploratory investigation of the pharmacokinetics of the drug administered through the dosage of hormones in serum LNG and EE2 for 28 days. | PK: 1 (0, 1, 2, 3, 4, 5, 6, 12 e 18 hours after administration), 2, 7, 14, 21 and 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Frederico, PI, Principal Investigator — LAL Clinica Pesquisa e Desenvolvimento Ltda
Locations (1):
- LAL Clínica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The study data will be maked available after journal's approbation. The manuscript contained all of data it has been submitted.

REFERENCES:
- [Result] Twaddle NC, Churchwell MI, Newbold RR, Delclos KB, Doerge DR. Determination using liquid-chromatography-electrospray tandem mass spectroscopy of ethinylestradiol serum pharmacokinetics in adult Sprague-Dawley rats. J Chromatogr B Analyt Technol Biomed Life Sci. 2003 Aug 15;793(2):309-15. doi: 10.1016/s1570-0232(03)00331-3. PMID 12906905
- [Result] Benagiano G, Carrara S, Filippi V. Safety, efficacy and patient satisfaction with continuous daily administration of levonorgestrel/ethinylestradiol oral contraceptives. Patient Prefer Adherence. 2009 Nov 3;3:131-43. doi: 10.2147/ppa.s3692. PMID 19936155
- [Result] Crosignani PG, Testa G, Vegetti W, Parazzini F. Ovarian activity during regular oral contraceptive use. Contraception. 1996 Nov;54(5):271-3. doi: 10.1016/s0010-7824(96)00178-3. PMID 8934059
- [Result] van Heusden AM, Fauser BC. Activity of the pituitary-ovarian axis in the pill-free interval during use of low-dose combined oral contraceptives. Contraception. 1999 Apr;59(4):237-43. doi: 10.1016/s0010-7824(99)00025-6. PMID 10457868
- [Result] Rossmanith WG, Steffens D, Schramm G. A comparative randomized trial on the impact of two low-dose oral contraceptives on ovarian activity, cervical permeability, and endometrial receptivity. Contraception. 1997 Jul;56(1):23-30. doi: 10.1016/s0010-7824(97)00070-x. PMID 9306028
- [Result] Hemrika DJ, Slaats EH, Kennedy JC, de Vries Robles-Korsen TJ, Schoemaker J. Pulsatile luteinizing hormone patterns in long term oral contraceptive users. J Clin Endocrinol Metab. 1993 Aug;77(2):420-6. doi: 10.1210/jcem.77.2.8345046.
- [Result] Kroll R, Reape KZ, Margolis M. The efficacy and safety of a low-dose, 91-day, extended-regimen oral contraceptive with continuous ethinyl estradiol. Contraception. 2010 Jan;81(1):41-8. doi: 10.1016/j.contraception.2009.07.003. PMID 20004272